CLINICAL TRIAL: NCT04581876
Title: A Single-arm, Prospective Study to Evaluate the Safety and Efficacy and of the Combination of Raltitrexed for Injection and Nab-Paclitaxel as Second-line Therapy in Treating Patients With Advanced Pancreatic Cancer
Brief Title: The Safety and Efficacy of the Combination of Raltitrexed for Injection and Nab-Paclitaxel in Advanced Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xian-Jun Yu, Vice President, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPAC-24
Record Dates: First submitted 2020-06-30; First posted 2020-10-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Pancreatic Cancer; Chemotherapy Effect
Keywords: Advanced pancreatic cancer; raltitrexed for injection; nab-paclitaxel
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — raltitrexed; Injections; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- raltitrexed for injection + nab-paclitaxel (Experimental): Patients receive raltitrexed 2mg/m2 (iv, 15min) and nab-paclitaxel at 125 mg/m2 on day 1 and day 15, q4w. Treatment repeats every 4 weeks until the disease recurrence or unacceptable toxicity, death or begin a novel treatment.
  Interventions: Drug: raltitrexed for injection; Drug: nab-paclitaxel

INTERVENTIONS:
Drug: raltitrexed for injection — Patients receive raltitrexed 2mg/m2 (iv, 15min) on day 1 and day 15, q4w. Treatment repeats every 4 weeks until the disease recurrence or unacceptable toxicity, death or begin a novel treatment.
  Other Names: raltitrexed
Drug: nab-paclitaxel — Patients receive nab-paclitaxel at 125 mg/m2 on day 1 and day 15, q4w. Treatment repeats every 4 weeks until the disease recurrence or unacceptable toxicity, death or begin a novel treatment.
  Other Names: albumin-bound paclitaxel

SUMMARY:
The present study is intended to investigate the safety and efficacy of the patients with confirmed advanced pancreatic cancer after treating with the combination of raltitrexed for injection and nab-paclitaxel.

DETAILED DESCRIPTION:
Conditions: Advanced pancreatic cancer subjects which were prospectively to receive first-line chemotherapy.

Keywords: Advanced pancreatic cancer; paclitaxel liposome; S-1 Interventions: Drug: paclitaxel liposome; Drug:S-1 Phase: Phase IV Study Type: Interventional

Study Design:

Allocation: Non-randomized Endpoint Classification: Efficacy/ Safety Study Intervention Model: single arm Primary Purpose: Treatment MedlinePlus related topics: Cancer, Pancreatic Cancer Drug Information available for: paclitaxel liposome：paclitaxel liposome for injection S-1：Tegafur, Gimeracil and Oteracil Potassium Capsules

Primary Outcome Measures:

To evaluate the Progression Free Survival of patients with advanced pancreatic cancer after treated with paclitaxel liposome plus S-1.

Secondary Outcome Measures:

To evaluate the Overall Response Rate、overall survival、disease control rate、Quality of Life、adverse events of patients with advanced pancreatic cancer after treated with paclitaxel liposome plus S-1.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed content obtained prior to treatment;
2. The patients were confirmed as advanced pancreatic cancer by histopathology or cytology;
3. At least one measurable objective lesion was identified based on the RECIST 1.1 criteria;
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
5. The expected survival after surgery ≥3 months;
6. Subjects had good compliance, were able to undergo treatment and follow-up, and voluntarily followed the relevant regulations of this study;
7. No contraindications to the use of raltitrexed for injection and nab-paclitaxel;
8. Age ≥18 years and ≤75 years;
9. Subjects of child-bearing age must agree to take effective contraceptive measures during the study period; Serum or urine pregnancy tests must be negative for women of childbearing age 7 days before the start of chemotherapy, during the monthly treatment interval and after the last treatment;
10. Women must be non-lactating.

Exclusion Criteria:

1. The target disease has cerebral metastasis;
2. The medical history and complications, which may affect patients' ability to participate in the study and their safety during the study, or interfere with explanation of the study results, for example: severe cardiovascular and cerebrovascular diseases, uncontrolled diabetes, uncontrolled hypertension, uncontrolled infection, active peptic ulcer, etc.;
3. Dementia, altered mental state, or any mental illness that prevents understanding or informed consent or questionnaires;
4. History of allergy or hypersensitivity to any therapeutic ingredient;
5. Combined with other malignant tumors excepted pancreatic cancer within the first 5 years of admission, excepted cured basal cell or squamous cell carcinoma of the skin, local prostate cancer after radical surgery, ductal carcinoma in situ after radical surgery;
6. Subjects with peripheral neuropathy ≥2 according to CTCAE version 5.0;
7. Physical examination or laboratory examination results are abnormal;

   1. Hematological dysfunction is defined as: i) absolute neutrophil (ANC) count <1.5 × 109 / L; ii) platelet (PLT) count: <100 × 109 / L; iii) hemoglobin (Hb) level<90g / L;
   2. Hepatic abnormalities are defined as: i) total bilirubin (TBil) levels: >1.5 times the upper limit of normal (ULN); ii) aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels >2.5 times the ULN >5 times ULN if liver metastases are present;
   3. Definition of renal dysfunction: serum creatinine >1.5 times ULN, or calculated creatinine clearance <50ml / min;
   4. Definition of abnormal blood coagulation function: International Normalized Ratio (INR) >1.5 times of ULN, and prothrombin time (PT) or activated partial thromboplastin time (aPTT) >1.5 times of ULN, unless the subject is receiving anti-antibodies Coagulation treatment.
8. Hepatitis B surface antigen positive (HBsAg), and subjects with peripheral blood hepatitis B virus DNA (HBV-DNA) titer ≥1×103 copies / L; if HBsAg is positive, and peripheral blood HBV-DNA <1×103 copy number / L, if the researcher believes that the subject's chronic hepatitis B is in a stable phase and does not increase the risk of the subject, the subject is eligible for selection;
9. Hepatitis C virus (HCV) or human immunodeficiency virus (HIV) positive;
10. Patients who need to combine other anti-tumor drugs;
11. Participation in any trial drug treatment or another interventional clinical trial 30 days before screening period.
12. Other conditions that researchers not think to be suitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
objective response rate | up to 36 months
  To evaluate the objective response rate of patients with advanced pancreatic cancer after treated with raltitrexed for injection plus nab-paclitaxel as second-line therapy.
progression free survival | up to 36 months
  To evaluate progression free survival of patients with advanced pancreatic cancer after treated with raltitrexed for injection plus nab-paclitaxel as second-line therapy.

SECONDARY OUTCOMES:
overall survival | up to 36 months
  To evaluate the overall survival of patients with advanced pancreatic cancer after treated with raltitrexed for injection plus nab-paclitaxel as second-line therapy.
adverse events | up to 36 months
  To evaluate the adverse events of patients with advanced pancreatic cancer after treated with raltitrexed for injection plus nab-paclitaxel as second-line therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Jun Yu, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No